CLINICAL TRIAL: NCT04535557
Title: An Expanded Access Protocol for Mobocertinib in Refractory Non-Small Cell Lung Cancer Patients With EGFR exon20 Insertion Mutations
Brief Title: An Expanded Access Protocol for Mobocertinib in Refractory Non-small Cell Lung Cancer (NSCLC) Participants With Epidermal Growth Factor Receptor (EGFR) Exon20 Insertion Mutations
Status: Approved for marketing | Type: Expanded Access
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: Mobocertinib EAP; U1111-1257-1911 (Registry Identifier: WHO)
Record Dates: First submitted 2020-08-28; First posted 2020-09-02 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Drug Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — mobocertinib

INTERVENTIONS:
Drug: Mobocertinib 160 mg — Mobocertinib 160 mg, capsule, orally, once daily in 28-day treatment cycles for up to approximately 4 months.

SUMMARY:
The purpose of this study is to provide expanded compassionate use access to mobocertinib, in participants with locally advanced or metastatic NSCLC harboring EGFR in-frame exon 20 insertion mutations and who have received at least 1 prior line of therapy for locally advanced or metastatic disease.

DETAILED DESCRIPTION:
The drug being tested in this study is called mobocertinib. Mobocertinib is being tested to treat people who have NSCLC with EGFR exon-20 insertion mutations who have failed the current standard of care (SOC) have no approved treatment therapies. Participants will be treated with mobocertinib until they experience progressive disease (PD) that requires an alternate therapy in the opinion of the physician, intolerable toxicity, or another discontinuation criterion. Treatment may be continued after PD if, in the opinion of the physician, the participant continues to experience clinical benefit.

The study will enroll approximately 100 participants. Enrollment will be based on unsolicited participant requests. All participants will be assigned to receive-

• Mobocertinib 160 milligram (mg)

Dose interruptions or reductions (first dose reduction- 120 mg and second dose reduction- 80 mg) will be implemented for participants who experience treatment-related adverse events (TEAEs), based on the clinical judgment of the investigator.

This multi-center trial will be conducted in the United States. The overall time to participate in this expanded access study is 4 months. The follow-up period for survival begins at the end of treatment (up to 30 days past last dose) and continues until participant discontinues.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically or cytologically confirmed locally advanced (and not a candidate for definitive therapy) or metastatic NSCLC
2. Have a documented EGFR in-frame exon 20 insertion mutations
3. . Must have received at least 1 prior line of therapy for locally advanced or metastatic disease
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
5. Normal QT interval on screening electrocardiogram (ECG), defined as QT interval corrected Fridericia (QTcF) of less than or equal to (<=) 450 milliseconds (ms) in males or <=470 ms in females

Exclusion Criteria:

1. Received small-molecule anticancer therapy (including cytotoxic chemotherapy and investigational agents) <=14 days prior to first dose of mobocertinib (except for reversible EGFR tyrosine kinase inhibitors (TKIs) [that is, erlotinib or gefitinib], which are allowed up to 7 days prior to the first dose of mobocertinib)
2. Received radiotherapy <=14 days prior to the first dose of mobocertinib or has not recovered from radiotherapy-related toxicities. Palliative radiation administered outside the chest and brain, stereotactic radiosurgery (SRS), and stereotactic body radiotherapy are allowed up to 7 days prior to the first dose
3. Have known active brain metastases. Brain metastases are allowed if they have been treated with surgery and/or radiation
4. Have current spinal cord compression or leptomeningeal disease
5. Have significant, uncontrolled, or active cardiovascular disease, including, but not restricted to:

   * Myocardial infarction (MI);
   * Unstable angina;
   * Congestive heart failure (CHF);
   * Clinically significant arrhythmia;
   * Ventricular arrhythmia; or
   * Cerebrovascular accident;
   * Transient ischemic attack.
   * Cardiac ejection fraction less than (<) 50 percent (%) by echocardiogram or multigated acquisition (MUGA) scan.
6. Have prolonged QTcF interval, or being treated with medications known to be associated with the development of Torsades de Pointes
7. Have presence of diarrhea that can be related to anti-tumoral treatment (including EGFR TKI, immune therapy, chemotherapy, and investigational therapies)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.